CLINICAL TRIAL: NCT06161038
Title: Precision Medicine for Nociception, Sngception and Proprioception.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202302118RINA
Record Dates: First submitted 2023-12-05; First posted 2023-12-07 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Rehabilitation; Pain, Shoulder; Pain, Chronic; Idiopathic Scoliosis
Keywords: Sng / Pain; Precision medicine; Next generation sequencing; Proprioception; Prolotherapy
MeSH Terms: conditions — Shoulder Pain; Chronic Pain; Pain | interventions — Lasers; Ultrasonography; Ultrasonic Therapy; Prolotherapy

STUDY DESIGN:
Intervention Model Description: 1. Cohort A-Myofascial pain syndrome The eligible patients first received LLLT with a 685-nm wavelength and an output of 30 mW at energy densities of 8 J/cm2 at trigger point of upper trapezius muscle.
     Then, they are conveniently assigned into two groups (40 subjects in each group): A. therapeutic ultrasound group; B. prolotherapy group. The same physician (the principal investigator) injects all patients to avoid inter-physician variability.
     Rescue therapy (cross-over treatment): If the participant does not satisfy with their first round treatment and the improvement of VAS is less than 10, then they are eligible to receive the rescue therapy-the treatment in the other group.
  2. Cohort B-idiopathic scoliosis:
  The recruited patients receive evaluation for once only. The collected parameters include Cobb's angle, spine rotational angle, VAS-pain and VAS-sng (visual analogue scale), pain threshold, strength and tone of paraspinal muscle, and SF-36.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A-A.therapeutic ultrasound group (Active Comparator): 1. Participants: Age between 20-100 years old who diagnosed as myofascial pain syndrome patients and willing to receive treatment.
  2. Intervention: Group A (A) receives 1 MHz therapeutic ultrasound for 5 min at a frequency of 2-3 times per week at the painful upper trapezius muscle.
  Interventions: Device: LASER; Device: Ultrasound; Drug: Prolotherapy
- Cohort A-B.prolotherapy group (Active Comparator): 1. Participants: Age between 20-100 years old who diagnosed as myofascial pain syndrome patients and willing to receive treatment.
  2. Intervention: Group B receives hypertonic prolotherapy at perimysium of upper trapezius muscle. The injectant is 5ml 5% dextrose solution.
  Interventions: Device: LASER; Device: Ultrasound; Drug: Prolotherapy
- Cohort B (No Intervention): 1. Participants: Age between 13-65 years old who diagnosed as idiopathic scoliosis The diagnosis of scoliosis was confirmed by antero-posterior plain Xray with Cobbs angle larger than 10 degrees.
  2. Intervention: None

INTERVENTIONS:
Device: LASER — LLLT with a 685-nm wavelength and an output of 30 mW (BTL-5000 Laser, BTL, Stevenage, UK) at energy densities of 8 J/cm2 at trigger point of upper trapezius muscle.
  Arms: Cohort A-A.therapeutic ultrasound group; Cohort A-B.prolotherapy group
Device: Ultrasound — 1 MHz therapeutic ultrasound for 5 min at a frequency of 4-6 times two week at the painful upper trapezius muscle.
  Other Names: Therapeutic ultrasound
  Arms: Cohort A-A.therapeutic ultrasound group; Cohort A-B.prolotherapy group
Drug: Prolotherapy — Hypertonic prolotherapy at perimysium of upper trapezius muscle. The injectant is 5ml 5% dextrose solution.
  Other Names: Hypertonic prolotherapy
  Arms: Cohort A-A.therapeutic ultrasound group; Cohort A-B.prolotherapy group

SUMMARY:
Precision medicine is defined as "an emerging approach for disease treatment and prevention that takes into account individual variability in genes, environment, and lifestyle for each person" by the Precision Medicine Initiative.

Patients have different response to different treatment modalities, and sore/pain medicine is no exception. In our experience, low-level laser (LLL), ultrasound, and prolotherapy can reduce sore /pain through different genetic pathway. Whether the therapeutic effect is controlled by the genetic variants of those sore /pain related genes or not, is still in debate. The aims of this study are (1) To set up next generation sequencing (NGS)-based approach to find genetic variants which can determine the response of sng/pain treatment modalities and the phenotype of idiopathic scoliosis. (2) To find possible metabolomics and proteomic markers of sng/pain. (3) To determine the algorithm of precision medicine for sng/pain control via the genetic markers.

Investigators will recruit 80 myofascial pain participant and 80 idiopathic scoliosis participant from Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital Bei-Hu Branch in 2023 and 2025. The myofascial pain participant participants will receive LLL, ultrasound, and prolotherapy, and the therapeutic effect will be recorded. The clinical trial will evaluate the Sng / pain (VAS) and muscle tone of the idiopathic scoliosis participant. The blood and urine samples from the first, the second, and the third visits will be analyzed by next generation sequencing, and mass spectrometry to find the possible biomarker in 2024 and 2025. Investigators expect to develop the individualized treatment plan by means of these biomarkers. Hopefully, the results will be widely applied in the field of sore /pain medicine.

DETAILED DESCRIPTION:
Precision medicine is defined as "an emerging approach for disease treatment and prevention that takes into account individual variability in genes, environment, and lifestyle for each person" by the Precision Medicine Initiative.

Pain is defined as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage or described in terms of such damage" by the International Association for the Study of Pain (IASP).Traditionally, soreness, or sng, is also included as one of the pain sensation. Recently, the investigators defined sngception as acid and/or soreness sensation in the somatosensory system, and revealed that analgesia in muscle is through substance P and Tac1.

According to the clinical outcome, some patients responded to physical agents well, and some preferred injections. The genetic variants of the above-mentioned genes might be the determining factors of differential therapeutic effects. However, it took about 4-8 weeks for a patient to switch from one treatment option to another one. If the investigators can determine the optimal treatment modality by genetic biomarkers, the treatment course and total expanse will decrease a lot.

The investigators hypothesize that the genetic variants of the proposed genes (TRPV1, ASIC1a, ASIC3, Tac1, COMT, TCL1A, POMC, RGS4, ASIC2, ASIC4, TRPA1, NK1R, G2A, GPR4, OGR1, TDAG8, TASK1, TASK2, TASK3, TREK1, P2X2, P2X3, P2X5, TRPV4, KCNK1, NTSR1, NTSR2, CaV3.2, Nav1.1, Piezo1, and Piezo2, Runx3 or Egr3, endothelin converting enzyme-like 1 (ECEL1), myosin heavy chain genes MYH3 and MYH8, myosin-binding protein C gene, MYBPC1, and TNNI2, TNNT3 and TPM2 that encode the muscle regulatory proteins troponin I, troponin T and beta-tropomyosin) could be the prognostic biomarkers of sng/pain treatments or proprioceptive function.

1.Specific Aims

1. To set up next generation sequencing (NGS)-based approach to find genetic variants which can determine the response of sng/pain treatment modalities and the phenotype of idiopathic scoliosis.
2. To find possible metabolomics and proteomic markers of sng/pain.
3. To determine the algorithm of precision medicine for sng/pain control via the genetic markers.

2.In the past years, our team had some achievements to justify the search of genetic variants for development of a new sore/pain treatment algorithm.

1. Analgesia of LLLT is through TRPV1.
2. Analgesia by therapeutic ultrasound is through ASIC3.
3. Dextrose injection decreased chronic muscle pain through ASIC1a.
4. Biomarker for sng/pain in fibromyalgia.

3.Study design

(1) Participants from cohort A-Myofascial pain syndrome: The investigators will recruit 80 participant from National Taiwan University Hospital and its Branch hospital.

B. Clinical trail design:

1. After obtaining the informed consent, the basic demographic data, including age, gender, job, education level, and past medical history of eligible participant are collected.
2. The eligible participant first received LLLT with a 685-nm wavelength and an output of 30 mW at energy densities of 8 J/cm2 at trigger point of upper trapezius muscle. The pre- and post-treatment VAS-pain and VAS-sng are collected for LLLT phenotype determination, respectively.
3. Then, they are conveniently assigned into two groups (40 subjects in each group): A. therapeutic ultrasound group; B. prolotherapy group. Group A receives therapeutic ultrasound. Group B receives hypertonic prolotherapy at perimysium of upper trapezius muscle. No other medication or physical modality was given to avoid efficacy interference in both groups.
4. The recruited participant receive evaluation before and after injection, and 2-week after injection. The primary outcome is VAS-pain and VAS-sng. The secondary outcomes are pain threshold, muscle tone, and SF-36. Venous blood and urine samples were collected at first visit and 2-week visit, respectively. The buffy coat is separated after centrifugation, and stored as well. The urine samples were aliquoted and stored at -80 ºC in a locked freezer for future analysis.
5. Rescue therapy (cross-over treatment): If the participant does not satisfy with their first round treatment and the improvement of VAS is less than 10, then they are eligible to receive the rescue therapy-the treatment in the other group. And they will return to clinic for another 2 weeks. The outcome variables will be collected in the 3rd visit as well.

(2) Participants from cohort B-idiopathic scoliosis: The investigators will recruit 80 participant from National Taiwan University Hospital and its Branch hospital, and Taichung Veteran Hospital.

B. Clinical Trail design:

1. After obtaining the informed consent, the basic demographic data, including age, gender, job, education level, physical activity level, and past medical history of eligible participant are collected.
2. The recruited participant receive evaluation for once only. The collected parameters include Cobb's angle, spine rotational angle, VAS-pain and VAS-sng, strength and tone of paraspinal muscle, and SF-36. Venous blood and urine samples were also collected.

Data analyses will be performed as previously described. Briefly, the raw sequencing data will be aligned to the reference human genome (Feb. 2009, GRCh37/hg19) using BWA-MEM. The investigators will use Picard to perform necessary data conversion, sorting and indexing. The main variant calling process, for both single nucleotide variants and indels, will be operated with the GATK software package. Structural variants will also be identified. The investigators will apply ANNOVAR to appropriately annotate the genetic variants; this include at least gene annotation, amino acid change annotation, SIFT scores, PolyPhen2 score, dbSNP identifiers, 1000 Genome Project allele frequencies, gnomAD allele frequencies and ClinVar database with variant clinical significance. The investigators will then use IGV to view the mapping and annotation of sequences on a graphic interface.

The allele frequencies of variants of interest will be compared between different groups of participants. The investigators will look for possible rare variants with very strong effects (the single-gene model) as well as relatively common variants with moderate to strong effects (the complex phenotype model).

ELIGIBILITY:
Inclusion Criteria:

1.Cohort A:

(1) Age between 20-100 years old. (2) VAS>=30 or VAS>=30 at 4 kg pressure (3) Diagnosed as myofascial pain syndrome patients and willing to receive treatment (including LLLT, therapeutic ultrasound, and local dextrose injection therapy) 2. Cohort B:

1. Age between 13-65 years old.
2. Diagnosed as idiopathic scoliosis The diagnosis of scoliosis was confirmed by antero-posterior plain Xray with Cobbs angle larger than 10 degrees.

Exclusion Criteria:

1.Cohort A: Those having active infection, malignancy, and hematological diseases were excluded. The patients had received local injection at upper trapezius within 6 months are also excluded.

2.Cohort B:

1. Those having active infection, malignancy, and hematological diseases were excluded.
2. Those having specific etiologies of scoliosis, including congenital scoliosis due to malformation or faulty segmentation of the vertebrae and neuromuscular scoliosis due to muscular imbalance, syndromic scoliosis or degenerative scoliosis.
3. Pregnancy.

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline Visual Analogue Scale.
  Visual Analogue Scale (VAS) anchor the patient's mark, providing a range of scores from 0-100. score 0 means 'no pain' and score 100 means 'pain worst'. VAS have been recommended: no pain (0 point), mild pain(10-40 point), moderate pain (50-70 point ), and severe pain (80-100 point).
Visual Analogue Scale (VAS) | Only cohort A: Change from Baseline Visual Analogue Scale at 2 weeks.
  Visual Analogue Scale (VAS) anchor the patient's mark, providing a range of scores from 0-100. score 0 means 'no pain' and score 100 means 'pain worst'. VAS have been recommended: no pain (0 point), mild pain(10-40 point), moderate pain (50-70 point ), and severe pain (80-100 point).
Visual Analogue Scale (VAS) | Only cohort A: Change from Baseline Visual Analogue Scale at 4 weeks (if crossover)
  Visual Analogue Scale (VAS) anchor the patient's mark, providing a range of scores from 0-100. score 0 means 'no pain' and score 100 means 'pain worst'. VAS have been recommended: no pain (0 point), mild pain(10-40 point), moderate pain (50-70 point ), and severe pain (80-100 point).

SECONDARY OUTCOMES:
Myoton-Muscle tone | Cohort A: Baseline, week 2, week 4 (if crossover); Cohort B: Baseline
  Muscle tone means state of muscle tension, which unit is Natural oscillation frequency [Hz]. This higher or lower value meaning is uncertainty. The range was from 10 to 30 Hz.
Myoton- Dynamic stiffness | Cohort A: Baseline, week 2, week 4 (if crossover); Cohort B: Baseline
  Muscle tone means muscle biomechanical properties, which unit is N/m. This higher or lower value meaning is uncertainty. The range was from 100 to 600 Hz.
Pain thresholds | Cohort A: Baseline, week 2, week 4 (if crossover); Cohort B: Baseline
  The item evaluate by SBMEDIC Algometer. The investigators used a device to press the participant's upper trapezius muscle until the subject call "uncomfortable" and then recorded the value. The investigators catch mean by three times.
  Pain thresholds range from 0 to 800 Kpa. Low thresholds means higher pain sensitivity (Pain tolerance) or muscle inflammation.
SF-36 | Cohort A: Baseline, week 2, week 4 (if crossover); Cohort B: Baseline
  Quality of life (36-Item Short Form Survey)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Bei-Hu Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data doesn't shared with other researchers.

REFERENCES:
- [Background] Assaraf E, Blecher R, Heinemann-Yerushalmi L, Krief S, Carmel Vinestock R, Biton IE, Brumfeld V, Rotkopf R, Avisar E, Agar G, Zelzer E. Piezo2 expressed in proprioceptive neurons is essential for skeletal integrity. Nat Commun. 2020 Jun 23;11(1):3168. doi: 10.1038/s41467-020-16971-6. PMID 32576830
- [Background] Avrampou K, Pryce KD, Ramakrishnan A, Sakloth F, Gaspari S, Serafini RA, Mitsi V, Polizu C, Swartz C, Ligas B, Richards A, Shen L, Carr FB, Zachariou V. RGS4 Maintains Chronic Pain Symptoms in Rodent Models. J Neurosci. 2019 Oct 16;39(42):8291-8304. doi: 10.1523/JNEUROSCI.3154-18.2019. Epub 2019 Jul 15. PMID 31308097
- [Background] Chang KV, Wu WT, Han DS, Ozcakar L. Static and Dynamic Shoulder Imaging to Predict Initial Effectiveness and Recurrence After Ultrasound-Guided Subacromial Corticosteroid Injections. Arch Phys Med Rehabil. 2017 Oct;98(10):1984-1994. doi: 10.1016/j.apmr.2017.01.022. Epub 2017 Feb 27. PMID 28245972
- [Background] Cho CH, Lho YM, Ha E, Hwang I, Song KS, Min BW, Bae KC, Kim DH. Up-regulation of acid-sensing ion channels in the capsule of the joint in frozen shoulder. Bone Joint J. 2015 Jun;97-B(6):824-9. doi: 10.1302/0301-620X.97B6.35254. PMID 26033064
- [Background] Choi JH, Yarishkin O, Kim E, Bae Y, Kim A, Kim SC, Ryoo K, Cho CH, Hwang EM, Park JY. TWIK-1/TASK-3 heterodimeric channels contribute to the neurotensin-mediated excitation of hippocampal dentate gyrus granule cells. Exp Mol Med. 2018 Nov 12;50(11):1-13. doi: 10.1038/s12276-018-0172-4. PMID 30416196
- [Background] Collins FS, Varmus H. A new initiative on precision medicine. N Engl J Med. 2015 Feb 26;372(9):793-5. doi: 10.1056/NEJMp1500523. Epub 2015 Jan 30. PMID 25635347
- [Background] Coste B, Houge G, Murray MF, Stitziel N, Bandell M, Giovanni MA, Philippakis A, Hoischen A, Riemer G, Steen U, Steen VM, Mathur J, Cox J, Lebo M, Rehm H, Weiss ST, Wood JN, Maas RL, Sunyaev SR, Patapoutian A. Gain-of-function mutations in the mechanically activated ion channel PIEZO2 cause a subtype of Distal Arthrogryposis. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):4667-72. doi: 10.1073/pnas.1221400110. Epub 2013 Mar 4. PMID 23487782
- [Background] Genovese TJ, Mao JJ. Genetic Predictors of Response to Acupuncture for Aromatase Inhibitor-Associated Arthralgia Among Breast Cancer Survivors. Pain Med. 2019 Jan 1;20(1):191-194. doi: 10.1093/pm/pny067. PMID 29912452
- [Background] Hsiung YC, Lin PC, Chen CS, Tung YC, Yang WS, Chen PL, Su TC. Identification of a novel LDLR disease-causing variant using capture-based next-generation sequencing screening of familial hypercholesterolemia patients in Taiwan. Atherosclerosis. 2018 Oct;277:440-447. doi: 10.1016/j.atherosclerosis.2018.08.022. PMID 30270083
- [Background] Li L, Wang HM, Shen Y. Chinese SF-36 Health Survey: translation, cultural adaptation, validation, and normalisation. J Epidemiol Community Health. 2003 Apr;57(4):259-63. doi: 10.1136/jech.57.4.259. PMID 12646540
- [Background] Liao HW, Kuo CH, Chao HC, Chen GY. Post-column infused internal standard assisted lipidomics profiling strategy and its application on phosphatidylcholine research. J Pharm Biomed Anal. 2020 Jan 30;178:112956. doi: 10.1016/j.jpba.2019.112956. Epub 2019 Oct 30. PMID 31704131
- [Background] Lin JH, Hung CH, Han DS, Chen ST, Lee CH, Sun WZ, Chen CC. Sensing acidosis: nociception or sngception? J Biomed Sci. 2018 Nov 29;25(1):85. doi: 10.1186/s12929-018-0486-5. PMID 30486810
- [Background] Lin YH, Wu CC, Lin YH, Lu YC, Chen CS, Liu TC, Chen PL, Hsu CJ. Targeted Next-Generation Sequencing Facilitates Genetic Diagnosis and Provides Novel Pathogenetic Insights into Deafness with Enlarged Vestibular Aqueduct. J Mol Diagn. 2019 Jan;21(1):138-148. doi: 10.1016/j.jmoldx.2018.08.007. Epub 2018 Sep 28. PMID 30268946
- [Background] Masingue M, Faure J, Sole G, Stojkovic T, Leonard-Louis S. A novel nonsense PIEZO2 mutation in a family with scoliosis and proprioceptive defect. Neuromuscul Disord. 2019 Jan;29(1):75-79. doi: 10.1016/j.nmd.2018.10.005. Epub 2018 Nov 8. PMID 30578100
- [Background] Niculescu AB, Le-Niculescu H, Levey DF, Roseberry K, Soe KC, Rogers J, Khan F, Jones T, Judd S, McCormick MA, Wessel AR, Williams A, Kurian SM, White FA. Towards precision medicine for pain: diagnostic biomarkers and repurposed drugs. Mol Psychiatry. 2019 Apr;24(4):501-522. doi: 10.1038/s41380-018-0345-5. Epub 2019 Feb 12. PMID 30755720
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Trobisch P, Suess O, Schwab F. Idiopathic scoliosis. Dtsch Arztebl Int. 2010 Dec;107(49):875-83; quiz 884. doi: 10.3238/arztebl.2010.0875. Epub 2010 Dec 10. PMID 21191550
- [Result] Cheng YR, Jiang BY, Chen CC. Acid-sensing ion channels: dual function proteins for chemo-sensing and mechano-sensing. J Biomed Sci. 2018 May 24;25(1):46. doi: 10.1186/s12929-018-0448-y. PMID 29793480
- [Result] Han DS, Lee CH, Shieh YD, Chen CC. Involvement of Substance P in the Analgesic Effect of Low-Level Laser Therapy in a Mouse Model of Chronic Widespread Muscle Pain. Pain Med. 2019 Oct 1;20(10):1963-1970. doi: 10.1093/pm/pnz056. PMID 30908578
- [Result] Hsu WH, Han DS, Ku WC, Chao YM, Chen CC, Lin YL. Metabolomic and proteomic characterization of sng and pain phenotypes in fibromyalgia. Eur J Pain. 2022 Feb;26(2):445-462. doi: 10.1002/ejp.1871. Epub 2021 Oct 26. PMID 34608709
- [Result] Hsu WH, Lee CH, Chao YM, Kuo CH, Ku WC, Chen CC, Lin YL. ASIC3-dependent metabolomics profiling of serum and urine in a mouse model of fibromyalgia. Sci Rep. 2019 Aug 20;9(1):12123. doi: 10.1038/s41598-019-48315-w. PMID 31431652